CLINICAL TRIAL: NCT02193945
Title: OZONE: Ocriplasmin Ellipsoid Zone Retrospective Data Collection Study
Brief Title: A Retrospective Chart Review of Patients Treated With Ocriplasmin for Symptomatic VMA
Acronym: OZONE
Status: Completed | Type: Observational
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Other Study IDs: TG-MV-022
Record Dates: First submitted 2014-07-11; First posted 2014-07-18 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Symptomatic Vitreomacular Adhesion (VMA)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to retrospectively review and further characterize anatomic and symptomatic changes over six months immediately following treatment of symptomatic vitreomacular adhesion (VMA) with JETREA® (ocriplasmin), including incidence, time to onset and resolution of anatomy and symptoms.

DETAILED DESCRIPTION:
This study (TG-MV-022) is a retrospective study utilizing Spectral-domain optical coherence tomography (SD-OCT) in patients treated previously with JETREA® for VMA. The objectives of this study are to retrospectively review and further characterize anatomic and symptomatic changes over six months immediately following treatment of VMA with JETREA® (ocriplasmin), including incidence, time to onset and resolution of anatomy and symptoms. The retrospective study will collect Heidelberg Spectralis® SD-OCT images which will be masked and uploaded to a Central Reading Center (CRC) for review and analysis. The CRC will evaluate anatomic endpoints of interest from both baseline optical coherence tomography (OCT) images and all follow-up OCT scans over the 6 month follow up period. Endpoints of interest include ellipsoid zone disruption, development of subretinal fluid, resolution of VMA and macular hole changes. Further, trained clinical personnel at the participating centers will transcribe data from the patients' records, to be entered into the study database.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age or older.
2. Have been treated with JETREA® for vitreomacular adhesion (VMA) between April 1, 2013 and December 31, 2013 with at least six months of follow up visits post injection. Note: If a patient's second eye was treated, only the first eye treated is eligible for study participation.
3. Have been imaged with Heidelberg Spectralis SD-OCT at least one time within 30 days prior to JETREA® injection.
4. Have been imaged with Heidelberg Spectralis SD-OCT at least two times post JETREA® injection with at least one scan between Days 1-21 and the second scan within six months,, including a corresponding visual acuity (VA).
5. Be willing and able to provide informed consent.

Exclusion Criteria:

1. Patients treated with JETREA® for medical conditions outside of the product label.
2. Patients with other retinal conditions that affect the vitreo-retinal interface, or can lead to retinal atrophy, including but not limited to:

   * Neovascular age-related macular degeneration;
   * Fibrovascular scar;
   * Diabetic macular edema; and
   * Proliferative diabetic retinopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been treated with JETREA® for Symptomatic vitreomacular adhesion (VMA)
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with ellipsoid zone disruption by Day 21 post-JETREA® injection, determined by a Central Reading Center (CRC), that was not present at baseline. | Day 21

SECONDARY OUTCOMES:
Proportion of patients with ellipsoid zone disruption, not present at baseline | Up to 6 months
Proportion of patients with ellipsoid zone disruption with resolution | Up to 6 months
Time to onset of ellipsoid zone disruption | Up to 6 months
Time to resolution of ellipsoid zone disruption | Up to 6 months
Proportion of patients that developed subretinal fluid, not present at baseline | Up to 6 months
Proportion of patients that developed subretinal fluid with resolution | Up to 6 months
Time to onset of subretinal fluid | Up to 6 months
Time to resolution of subretinal fluid | Up to 6 months
Proportion of patients with nonsurgical resolution of VMA by Day 28 | Day 28
Time to resolution of VMA | Up to 6 months
Proportion of patients that developed a macular hole by Day 28, not present at baseline | Day 28
Proportion of patients with nonsurgical closure of macular hole, if present at baseline by Day 28 | Day 28
Proportion of patients with worsening (enlargement) of macular hole, if present at baseline | Up to 6 months
No change of macular hole, if present at baseline | Up to 6 months
Proportion of patients that underwent vitrectomy | Up to 6 months
Visual Acuity (VA) changes from baseline | Up to 6 months
Other findings as examined and documented in the patient's medical records | Up to 6 months
  * Impaired pupillary reflex
  * Dyschromatopsia
  * ERG changes
  * Vascular changes
  * Visual field constriction
  * Lens changes post- JETREA® injection including, subluxation, dislocation, phacodenesis
  * Other changes in quality of vision including, darkness of vision, dark adaptation changes
Monitoring of Adverse Drug Reactions (ADRs) | Up to 6 motnths

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Retinal Diagnostic Center, Campbell, California
  - Scripps Clinic, La Jolla, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Marietta Eye Clinic, Marietta, Georgia
  - Rush university medical center-Dept ophthalmology, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Sabates Eye Centers, Leawood, Kansas
  - Carl W. Baker, Paducah, Kentucky
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - Sierra Eye Associates, Reno, Nevada
  - Eyesight Ophthalmic Services, Portsmouth, New Hampshire
  - MaculaCare, New York, New York
  - Duke University Eye Center, Durham, North Carolina
  - Wills Eye Institute, Philadelphia, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates, P.C., Kingsport, Tennessee
  - Retina Consultants of Houston, Houston, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Retina Specialists, Plano, Texas
  - Retina Associates of Utah, P.C., Salt Lake City, Utah
  - West Virginia University Eye Institute, Morgantown, West Virginia